CLINICAL TRIAL: NCT01001559
Title: Combination Deplin® and Antidepressant Therapy Compared to Antidepressant Therapy Alone for an Episode of Major Depression- a Retrospective Analysis
Brief Title: Combination Deplin® and Antidepressant Therapy for a Major Depressive Episode (MDE)- a Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Pamlab, Inc. (Industry)
Collaborators: Red Oak Psychiatry Associates, PA (Unknown); Baylor Health Care System (Other)
Responsible Party: Sponsor
Other Study IDs: Pamlab D-005
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-11

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Combination therapy; antidepressant; Deplin; folate; methylfolate
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — 5-methyltetrahydrofolate; Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Deplin + antidepressant: Deplin in combination with a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI)
  Interventions: Drug: L-methylfolate; Drug: Selective serotonin reuptake inhibitor (SSRI); Drug: Serotonin and norepinephrine reuptake inhibitor (SNRI)
- Antidepressant alone: SSRI or SNRI alone
  Interventions: Drug: Selective serotonin reuptake inhibitor (SSRI); Drug: Serotonin and norepinephrine reuptake inhibitor (SNRI)

INTERVENTIONS:
Drug: L-methylfolate — Subjects must have been on their respective therapies for a minimum of 60 days. L-methylfolate dosing was 7.5 mg or 15 mg daily
  Other Names: Deplin
  Groups: Deplin + antidepressant
Drug: Selective serotonin reuptake inhibitor (SSRI) — Subject must have been on their respective therapy for a minimum of 60 days. Because this was an observational retrospective analysis, dosing of SSRI/SNRI varied on a per patient basis.
Drug: Serotonin and norepinephrine reuptake inhibitor (SNRI) — Subject must have been on their respective therapy for a minimum of 60 days. Because this was an observational retrospective analysis, dosing of SSRI/SNRI varied on a per patient basis.

SUMMARY:
This is a retrospective chart review study to determine if Deplin® 7.5mg-15mg combined with an antidepressant is better than an antidepressant alone in adults with major depression.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18-70
* The active arm (Arm #1) includes randomly selected 100-125 charts of patients with a primary diagnosis of major depression and a CGI-S of ≥4 who began Deplin and SSRI or SNRI therapy at the same time beginning in January 2007 to the present; and, Control group (Arm #2) includes randomly selected 125-150 charts of patients with a primary diagnosis of major depression who began SSRI or SNRI therapy matched in severity (CGI-S of ≥4)

Exclusion Criteria:

* Folic acid >400 mcg taken at any time during the study
* Psychotic features in the current episode or a history of psychotic features
* Any bipolar disorder (current or past) or any psychotic disorder (current or past)
* Current or past treatment with vagus nerve stimulation, ECT, or transcranial magnetic stimulation
* Antipsychotic therapy in conjunction with their antidepressant currently or in past 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ages 18-70 experiencing an episode of major depression
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence D Ginsberg, MD, Principal Investigator — Red Oak Psychiatry Associates, PA
Locations (1):
- Red Oak Psychiatry Associates, PA, Houston, Texas, United States

REFERENCES:
- [Result] Ginsberg LD, Oubre AY, Daoud YA. L-methylfolate Plus SSRI or SNRI from Treatment Initiation Compared to SSRI or SNRI Monotherapy in a Major Depressive Episode. Innov Clin Neurosci. 2011 Jan;8(1):19-28. PMID 21311704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single site, retrospective chart review of subjects administered a combination of Deplin and an SSRI or SNRI. The 242 subjects were 18-70 years of age (inclusive) and received their respective therapies between January 2007 and September 2009.
Pre-assignment Details: Criteria that excluded patients were folic acid supplementation >400mcg, current or a history of psychotic features, bipolar disorder, a history of vagus nerve stimulation, electroconvulsive, or transcranial magnetic stimulation therapy. Any concomitant antipsychotic therapy in the most recent 4 weeks.
Period: Overall Study
Arm/Group | Deplin + Antidepressant | Antidepressant Alone
Started | 95 | 147
Completed | 95 | 147
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deplin + Antidepressant | Antidepressant Alone | Total
Number analyzed (Participants) | 95 | 147 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (11.9) | 41.4 (11.7) | 43.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 98 | 160
  Male | 33 | 49 | 82

OUTCOME MEASURES:

1. Primary Outcome: Improvement as Measured by Change in Clinical Global Impression of Severity (CGI-S) Rating From Baseline
Description: The Clinical Global Impression of Severity (CGI-S) Rating evaluates the severity of individual symptoms and treatment response in patients with mental disorders. The CGI-S is a 7-point scale that that requires the clinician to rate the severity of the patient's illness at the time of assessment. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms.
  Number of patients with an improvement in CGI-S scores as demonstrated by a reduction in ≥2 points (major improvement) from baseline.
Time Frame: 60 days
Population: All participants
Measure: Number; unit: Participants
Arm/Group | Deplin + Antidepressant | Antidepressant Alone
Number analyzed (Participants) | 95 | 147
Participants | 17 | 10

2. Secondary Outcome: Length of Time to Peak Response, as Determined by the Clinical Global Impression of Severity (CGI-S) Scale
Description: The Clinical Global Impression of Severity (CGI-S) Rating evaluates the severity of individual symptoms and treatment response in patients with mental disorders. The CGI-S is a 7-point scale that that requires the clinician to rate the severity of the patient's illness at the time of assessment. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms.
  Median times to peak response. Peak response defined as the first improvement of two or more in the CGI-S from initial visit, and measured the time to the occurrence.
Time Frame: 60 days
Population: All participants
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Deplin + Antidepressant | Antidepressant Alone
Number analyzed (Participants) | 95 | 147
Days | 177 [85 to 299] | 231 [126 to 540]

3. Secondary Outcome: Number of Hospitalizations Due to MDD
Description: Number of hospitalizations due to MDD during treatment were assessed during this retrospective analysis of L-methylfolate plus SSRI/SNRI at treatment initiation (n=95) and SSRI/SNRI monotherapy (n-147) from patient charts
Time Frame: 60 days
Measure: Number; unit: Hospitalizations due to MDD
Arm/Group | Deplin + Antidepressant | Antidepressant Alone
Number analyzed (Participants) | 95 | 147
Hospitalizations due to MDD | 1 | 4

4. Secondary Outcome: Absolute Count of Alterations in Therapy Required, Such as Dose Increases, Antidepressant Substitutions, or Addition of Augmentation Medications
Time Frame: 60 days
Measure: Number; unit: Alterations in antidepressant therapy
Arm/Group | Deplin + Antidepressant | Antidepressant Alone
Number analyzed (Participants) | 95 | 147
Alterations in antidepressant therapy | 135 | 263

ADVERSE EVENTS:
Time Frame: AE reporting occurred between January 2007 and September 2009
Arm/Group | Deplin + Antidepressant | Antidepressant Alone
Serious Adverse Events (participants affected / at risk) | 1/93 | 3/103
Other Adverse Events (participants affected / at risk) | 56/93 | 68/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deplin + Antidepressant (N=93) | Antidepressant Alone (N=103)
Hospitalization (General disorders) | 1 (1) | 3 (3) — Limited information regarding SAEs is available. Four hospitalizations, among three subjects in the Antidepressant Alone arm, and one hospitalization in the Deplin + Antidepressant arm occurred. No information regarding AE term or SOC is available.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deplin + Antidepressant (N=93) | Antidepressant Alone (N=103)
Sexual Dysfunction (Reproductive system and breast disorders) | 11 (11) | 15 (15)
Somnolence (Nervous system disorders) | 12 (12) | 12 (12)
Nausea (Gastrointestinal disorders) | 9 (9) | 9 (9)
Dizziness (Nervous system disorders) | 3 (3) | 7 (7)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (6)
Agitation (Psychiatric disorders) | 3 (3) | 6 (6)
Decreased Appetite (Psychiatric disorders) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (7) | 4 (4)
Fatigue (General disorders) | 5 (5) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No